CLINICAL TRIAL: NCT00913796
Title: Metabolic Acidosis and Its Impact on Mineral Metabolism and Physical Performance in Renal Transplant Patients
Brief Title: Metabolic Acidosis in Renal Transplant Patients
Acronym: MART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Texas Southwestern Medical Center (Other); Swiss Federal Institute of Technology (Other)
Responsible Party: Prof. Dr. Patrice Max Ambühl, University Hospital Zurich
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3200B0-112299
Record Dates: First submitted 2009-04-01; First posted 2009-06-04 (Estimated); Last update posted 2010-10-22 (Estimated); Status verified 2009-06

CONDITIONS: Renal Transplant Patients; Metabolic Acidosis; Physical Capacity; Bone Disease; Mineral Metabolism
Keywords: Renal transplantation; Metabolic acidosis; Physical capacity; Bone histology; Bone histomorphometry; Parathyroid function; Calcium and phosphate metabolism
MeSH Terms: conditions — Acidosis; Bone Diseases | interventions — Potassium Citrate; Potassium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Postassium citrate (Experimental): Aim: correction of metabolic acidosis
  Interventions: Drug: Potassium citrate
- Potassium chloride (Active Comparator): Potassium chloride is given to compensate for any possible effects of potassium in potassium citrate (primary treatment).
  Interventions: Drug: Potassium chloride

INTERVENTIONS:
Drug: Potassium citrate — 2.41 gram of citrate b.i.d. for 12 months. Dosage to be adjusted according to serum potassium concentration.
  Arms: Postassium citrate
Drug: Potassium chloride — 370 mg potassium t.i.d. for 12 months. Dosage to be adjusted according to serum postassium concentration.
  Arms: Potassium chloride

SUMMARY:
Acidosis (accumulation of acid in the body) may be an underrecognized problem in patients after renal transplantation. It may have consequences on physical performance due to negative effects on bone and muscle metabolism.

Therefore, the purpose of this study is

1. to determine the status of physical capacity and bone structure in renal transplant patients with metabolic acidosis
2. to study the effect of substituting base equivalents (citrate) on acid/base status of renal transplant patients with acidosis
3. to compare the status of physical capacity and bone structure in renal transplant patients with metabolic acidosis before and after substitution with citrate

DETAILED DESCRIPTION:
Chronic kidney disease is developing to become one of the major health problems in the Western world with more than one million patients on renal replacement therapy, and many more expected in the years ahead [1]. Survival of patients with end stage renal disease has become possible with the introduction of dialysis therapy. Renal transplantation has resulted both in further reduction of mortality and improvement in quality of life for patients with end stage renal disease. Nevertheless, successful transplantation with regard to graft and patient survival is still associated with significant morbidity. Apart from infectious complications and cardiovascular disease, limitations in physical capacity from musculoskeletal disorders have become a relevant problem, resulting in reduced quality of life, poor physical functioning and inability to work.

Muscle and bone metabolism in chronic kidney disease are typically disturbed resulting in significant pathology and dysfunction of the affected tissues. They are associated with metabolic disorders related to renal insufficiency, among which metabolic acidosis is a major contributor. Metabolic acidosis is a well recognized problem in renal transplant patients. However, its prevalence, pathogenesis, course and sequelae are not well established. In particular, its relation to post-transplant bone and muscle disorders, and the impact on physical capabilities in renal transplant patients have not been comprehensively investigated so far.

The purpose of the proposed project is to examine the characteristics and pathogenesis of post-transplant metabolic acidosis, and its relation to bone and muscle pathologies and impact on physical capabilities in renal transplant patients. In particular, the following aims are proposed to investigate in de novo and long-term renal transplantation:

Aim # 1: To examine the type, degree and course of metabolic acidosis in renal transplant patients, early and long-term after transplantation

Aim # 2: To examine alterations in mineral and bone metabolism, and bone structure, and their relationship to the acid/base disorder

Aim # 3: To examine overall physical performance, exercise capacity and muscle energy content, and their relationship to the acid/base disorder

In order to analyze secondary effects of subclinical and overt acidosis on bone (Aim # 2) and muscle (Aim # 3), patients will be studied at baseline, and then be supplemented with base equivalents in order to achieve a stable plasma serum bicarbonate concentration of 24-26 mmol/l, and be reexamined thereafter. Completion of the three aims will allow to comprehensively analyze the pathogenesis of and interrelations between acid/base status, mineral metabolism, bone disorders and muscle function in renal transplant patients. This will be the first study to link metabolic alterations to structural and functional measures of the musculoskeletal system, and to the impact of the resulting pathologies on physical disabilities in patients with a kidney graft. We are in dire need to know the magnitude of the problem, whether to treat, and how aggressive to treat these patients. The results of this project will be indispensable regarding justification to rigorously evaluate and treat metabolic acidosis in patients with chronic renal insufficiency and after transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a renal graft having been transplanted within the previous 8 years and being at least 3 months post transplantation, or, patients scheduled to undergo transplantation from a living organ donor within the upcoming 3 months
* Venous serum bicarbonate concentration < 24 mmol/L at time of baseline determination
* Renal transplant function with a calculated glomerular filtration rate (GFR) greater or equal 30 ml/min according to the Cockcroft-Gault formula
* Immunosuppressive therapy including a calcineurin inhibitor (cyclosporine A or tacrolimus)
* Age 20 through 65 years of either sex
* Written informed consent for study participation

Exclusion Criteria:

* Acute rejection episode requiring specific therapy within 4 weeks before study inclusion
* Severe impairment in general health and/or physical handicaps (malignant neoplasia, catabolic state, acute systemic infection requiring therapy)
* Mental illness, psychiatric disorder
* Tetracycline intolerance
* Planned or "overt" pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2007-12; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Correction of metabolic acidosis | 12 months

SECONDARY OUTCOMES:
Improvement in physical capacity | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrice M. Ambühl, M.D., Principal Investigator — University of Zurich
Locations (1):
- University Hospital of Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Starke A, Corsenca A, Kohler T, Knubben J, Kraenzlin M, Uebelhart D, Wuthrich RP, von Rechenberg B, Muller R, Ambuhl PM. Correction of metabolic acidosis with potassium citrate in renal transplant patients and its effect on bone quality. Clin J Am Soc Nephrol. 2012 Sep;7(9):1461-72. doi: 10.2215/CJN.01100112. Epub 2012 Jul 5. PMID 22773591